CLINICAL TRIAL: NCT00503165
Title: A Phase IV, Single Group Study to Evaluate the Immunogenicity and Safety in UK Laboratory Workers of a Licensed Hib and Meningococcal C Conjugate Combined Vaccine (Menitorix)
Brief Title: A Phase IV Study to Evaluate the Immunogenicity and Safety in UK Laboratory Workers of Menitorix
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Public Health England (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: StaMen
Record Dates: First submitted 2007-07-17; First posted 2007-07-18 (Estimated); Last update posted 2019-03-22 (Actual); Status verified 2008-02

CONDITIONS: Vaccination
Keywords: Menitorix; vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: Menitorix (MenC and Hib conjugate)

SUMMARY:
Menitorix is a combined Hib conjugate and meningococcal C conjugate vaccine made by GlaxoSmithKline. It is currently licensed and recommended as a booster vaccination for UK children in the second year of life.

It is important that staff who have a potential occupational exposure to infectious disease are afforded protection where possible. The licensure and availability of Menitorix provides the opportunity to vaccinate such staff.

Immune responses that are indicative of protection have been established for both Hib and meningococcal C disease. It is therefore proposed that the immune responses of those laboratory staff taking part be measured as data currently available following Menitorix vaccination is in naïve children and adults. This study will also allow us to provide occupational healthcare to laboratory workers.

Participation in the study would be offered to all those staff considered to be at occupational health risk of Hib or meningococcal C disease at the Manchester HPA site. This will be a single group study in that everyone enrolled will receive a single dose of Menitorix and will have blood collected prior to and 4-6 weeks following vaccination.

Assessment of whether protective levels of antibody have been achieved will be made using the blood sample taken 4-6 weeks after vaccination. Extra dose(s) will be offered to any subjects whose levels are not considered to confer protection as described later in this protocol. Subjects receiving and extra vaccination will be offered and a further blood test 4-6 weeks later to allow antibody levels to be checked again.

DETAILED DESCRIPTION:
Menitorix is a combined Hib conjugate and meningococcal C conjugate vaccine made by GlaxoSmithKline. It is currently licensed and recommended as a booster vaccination for UK children in the second year of life.

It is important that staff who have a potential occupational exposure to infectious disease are afforded protection where possible [HPA Occupational Health Policy [Appendix 1]; HSE Safe working and the prevention of infection in clinical laboratories and similar facilities, 2003]. The licensure and availability of Menitorix provides the opportunity to vaccinate such staff.

Immune responses that are indicative of protection have been established for both Hib and meningococcal C disease [Andrews et al., 2003; Kayhty et al., 1983]. It is therefore proposed that the immune responses of those laboratory staff taking part be measured as data currently available following Menitorix vaccination is in naïve children and adults [Tejedor et al., 2006a and b; Carmona et al., 2006; Habermehl et al., 2006; Pace et al., 2006]. This study will also allow us to provide occupational healthcare to laboratory workers.

Laboratory staff at Manchester have not received a Hib vaccine although they have received a number of meningococcal vaccines with the majority having received their meningococcal serogroup C conjugate vaccine in 1999. Certain staff would have received bivalent meningococcal A and C prior to the conjugate vaccine which has recently been demonstrated to hinder the induction of immunological memory by the conjugate vaccine [Vu et al., 2006]. Following the conjugate vaccine many staff have since received a quadrivalent A/C/Y/W135 polysaccharide vaccine in the following seven years, but little is known about the duration of protection in this age group.

Receiving a polysaccharide vaccine following a conjugate does induce an elevated antibody response but it is known that polysaccharide vaccination does not generate memory B cells and can result in the loss of the ability to mount subsequent memory antibody responses, as was observed by MacLennan et al. for Neisseria meningitidis group C anticapsular antibody responses [MacLennan et al., 2001]. The clinical importance of loss of immunological memory or induction of antibody hyporesponsiveness, is unknown. However, in addition to dampening antibody responses to a subsequent immunisation, a delay or impaired serum antibody response upon encountering an encapsulated pathogen could theoretically increase susceptibility to developing disease. Such a mechanism may explain the higher rate of otitis media observed after administration of 23-valent pneumococcal polysaccharide vaccine to Dutch children primed with a 7-valent pneumococcal polysaccharide protein conjugate vaccine as compared with the rate in controls given hepatitis B vaccine (P=0.0001) [Veenhoven et al., 2003]. In contrast, during the six months between the conjugate vaccination and booster there was a trend in favor of fewer episodes of otitis in the pneumococcal-vaccinated group.

It appears that staff will benefit from both the Hib and serogroup C conjugate vaccinations.

Assessments in this study:

Participation in the study would be offered to all those staff considered to be at occupational health risk of Hib or meningococcal C disease at the Manchester HPA site. The maximum number of participants would therefore be 30. This will be a single group study in that everyone enrolled will receive a single dose of Menitorix and will have blood collected prior to and 4-6 weeks following vaccination.

Local anaesthetic cream will be offered to minimise discomfort of the blood tests and fully trained staff will carry out all procedures.

Assessment of whether protective levels of antibody have been achieved will be made using the blood sample taken 4-6 weeks after vaccination. Extra dose(s) will be offered to any subjects whose levels are not considered to confer protection as described later in this protocol. Subjects receiving and extra vaccination will be offered and a further blood test 4-6 weeks later to allow antibody levels to be checked again.

Samples will be sent to collaborating laboratories of the National Vaccine Evaluation Consortium for assessment of responses to vaccinations.

ELIGIBILITY:
Inclusion Criteria:

* No contraindications to vaccination as specified in the "Green Book" - Immunisation Against Infectious Disease, HMSO.
* Written informed consent

Exclusion Criteria:

* Known or suspected pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2007-07; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Determine serum bactericidal antibody levels against Neisseria meningitis serogroup C. | 1 month after vaccination

SECONDARY OUTCOMES:
Determine anti-Hib IgG concentration (ELISA) | 1 month after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Ed Kaczmarski, MBBS, Principal Investigator — Public Health England
Locations (1):
- Health Protection Agency, Manchester Laboratory., Manchester, United Kingdom

REFERENCES:
- [Background] Findlow J, Findlow H, Frankland S, Holland A, Holme D, Newton E, Southern J, Waight P, Kaczmarski E, Miller E, Borrow R. Evaluation of the safety and immunogenicity in United Kingdom laboratory workers of a combined Haemophilus influenzae type b and meningococcal capsular group C conjugate vaccine. J Occup Med Toxicol. 2014 Jul 16;9:26. doi: 10.1186/1745-6673-9-26. eCollection 2014. PMID 25071861
- See also: Published study results — https://www.ncbi.nlm.nih.gov/pubmed/25071861